CLINICAL TRIAL: NCT03945396
Title: Efficacy of a Multidisciplinary Intervention and Homeopahy for Overweight or Obesity in Mexican Adolescents: a Study Protocol for a Randomized Double-blind, Placebo-controlled Trial
Brief Title: Homeopathy for Overweight and Obesity in Mexican Adolescents
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Emma del Carmen Macías-Cortés, MD, PhD, Head of homeopathy outpatient service, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HJM 0572/19-1
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Overweight; Homeopathy; Calcarea carbonica ostrearum; Mexico
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, double-blind, parallel, superiority trial with 3 month study duration.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary intervention + homeopathic medication (Experimental): Multidisciplinary intervention (diet, exercise program, motivational support) and Calcarea carbonica ostrearum 30c.
  A single dose of Calcarea carbonica ostrearum 30C dissolved in a 30 ml bottle of 30% alcohol-distilled water. Patients will receive 8 drops PO three times per day prior agitation.
  Interventions: Drug: Homeopathic Medication; Other: Multidisciplinary intervention (Exercise program, diet, motivational support)
- Multidisciplinary intervention + homeopathic placebo (Active Comparator): Multidisciplinary intervention (diet, exercise program, motivational support) and placebo.
  Placebo will be prepared with 30% alcohol-distilled water only, in the same 30 ml bottle. Patients will receive 8 drops PO three times per day prior agitation.
  Interventions: Other: Multidisciplinary intervention (Exercise program, diet, motivational support); Drug: Homeopathic placebo

INTERVENTIONS:
Drug: Homeopathic Medication — A homeopathic mineral medicine, form of impure calcium carbonate, CaCO3, which can be found in nature in different niches, from limestone to eggshells.
  Other Names: Calcarea carbonica ostrearum
  Arms: Multidisciplinary intervention + homeopathic medication
Other: Multidisciplinary intervention (Exercise program, diet, motivational support) — Exercise program: includes a five-times per week routine: warm-up during 10 to 15 minutes, then 40 minutes of aerobic exercise that will be increased progressively until reaching 60 minutes. Thereafter, muscular strength initiating 5%, and increasing until 10 to 15% of body weight. Then, 10 to 15 minutes of stretching. Finally, 5 min cool-down.
  Diet: Subjects will receive a balance diet calculated based on energetic needs according FAO: 15-20% of proteins, 50-60% of carbohydrate, 20-25% of fat per day.
  Motivational support: 50 min session where empathy and neutral understanding of the perspective and feelings of the adolescent, and his family, are fostered to motivate the change and to state realistic goals in reducing weight.
  Other Names: Combined dietary-behavioral-physical activity intervention
Drug: Homeopathic placebo — A 30 ml bottle of 30% alcohol-distilled water.
  Other Names: Placebo
  Arms: Multidisciplinary intervention + homeopathic placebo

SUMMARY:
This study evaluates the efficacy of a multidisciplinary intervention (diet, exercise, motivational support and homeopathy or placebo) for overweight and obesity in Mexican adolescents. Half of study participants will receive the multidisciplinary intervention plus Calcarea carbonica ostrearum, a homeopathic medicine, while the other half will receive the same multidisciplinary intervention plus placebo.

DETAILED DESCRIPTION:
Overweight and obesity in children and adolescents are a major public health issue in Mexico. Whilst many factors (genetic, cultural, socioeconomic and environmental) contribute to develop obesity during childhood, a multidisciplinary intervention (nutritional, behavioral and exercise) is the best approach to improve weight loss. In Mexico, the use of homeopathy for obesity is widespread. Although there are some homeopathic medicines used for obese individuals, there is a lack of well-designed clinical trials to demonstrate its efficacy in weight loss. Calcarea carbonica ostrearum is a homeopathic mineral medicine. Previously, it has been demonstrated that Calcarea carbonica has an effect in reducing the percentage of fat in adolescents.

Therefore, a randomized, placebo-controlled, double-blind, parallel, superiority trial with a 3 month study duration, will be conducted to prove the efficacy and safety of Calcarea carbonica ostrearum in reducing weight, body mass index (BMI) and fat percentage, as well as, to prove its effect on the lipid profile, fasting serum glucose, glycosylated hemoglobin and insulin.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 19 years old.
* At least elementary school.
* Overweight (BMI ≥ 85th but <95th percentile based on the Centers for Disease Control and Prevention growth chart) or obese (BMI ≥95th percentile).
* Fasting serum glucose <126 mg/dl.
* Glycosylated hemoglobin <6.5%.
* With symptoms that match with Calcarea carbonica ostrearum.
* Willingness to participate, and verbal and written consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Cases already undergoing treatment (homeopathic, nutritional or structured physical activity) for obesity within last three months.
* Currently use of metformin, orlistat, insulin, other antidiabetic medication, contraceptive pills, medications with effects on lipid metabolism [thiazide and loop diuretics, β and α receptor blockers, antiepileptic drugs (carbamazepine, phenytoin, valproic acid, phenobarbital), antipsychotics (clozapine), protease inhibitors (amprenavir, indinavir, nelfinavir, ritonavir, saquinavir), tamoxifen, raloxifene, isotretinoin, acitretin, ciclosporin, azathioprine, sirolimus].
* Any condition that prevents physical exercise.
* Diabetes, hypertension, thyroid diseases, Down syndrome, mental retardation.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean total weight in kilograms (kg) | At baseline and week 4, 8 and 12.
  Weight measured with the participants barefooted and lightly dressed, with a Tanita scale Fitscan BC-545 F segmental body composition monitor. The scale has an eight electrode body composition monitor that displays twenty readings; ten whole body and ten segmental (arms, legs and trunk area).
Change from baseline in percentage of body fat | At baseline and week 4, 8 and 12.
  Body fat measured with Tanita scale Fitscan BC-545 F segmental body composition monitor. Values greater than 30% for females, and 25% for males, are considered high and of risk

SECONDARY OUTCOMES:
Change from baseline in mean total body mass index (BMI). | At baseline and week 4, 8 and 12.
  Weight/height2 (kg/m2). Overweight (BMI ≥ 85th but <95th percentile based on the Centers for Disease Control and Prevention growth chart) or obese (BMI ≥95th percentile).
Change from baseline in mean total fat mass index | At baseline and week 4, 8 and 12.
  Calculated by dividing fat weight in kilograms by height in meters squared.
Change from baseline in mean total lean body mass (kg). | At baseline and week 4, 8 and 12.
  Calculated by subtracting body fat weight from total body weight: total body weight is lean plus fat
Change from baseline waist-hip ratio. | At baseline and week 4, 8 and 12.
  Calculated as waist measurement divided by hip measurement.
Change from baseline in mean total lean muscle mass (kg). | At baseline and week 4, 8 and 12.
  Calculated by total weight of the body minus all the weight due to the fat mass.
Number and severity of all adverse events | After participants consent and enrolled in the study and 15 days after study completion.
  Adverse event will be defined as any untoward medical occurrence in a subject without regard to the possibility of a causal relationship.

OTHER OUTCOMES:
Change from baseline in mean total fasting serum glucose (mg/dL) | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using an automated chemical analyzer (Advia®1200). Glucose will be assayed by the glucose-oxidase method.
Change from baseline in mean total fasting serum triglycerides (mg/dL) | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using an automated chemical analyzer (Advia®1200).
Change from baseline in mean total cholesterol (mg/dL) | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using an automated chemical analyzer (Advia®1200).
Change from baseline in mean total high-density cholesterol (mg/dL) | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using an automated chemical analyzer (Advia®1200).
Change from baseline in mean total low-density cholesterol (mg/dL) | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using an automated chemical analyzer (Advia®1200).
Change from baseline in percentage of glycosylated hemoglobin | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using an automated chemical analyzer (Advia®1200).
Change from baseline in mean total insulin (mU/ml) | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using a chemiluminescence technique (Immulite®2000TSH Third Generation).
Change from baseline in mean total thyroid-stimulating hormone (mU/L) | At baseline and week 12.
  Blood samples will be collected by venipuncture in the antecubital region of patients after 10-12 hours of overnight fasting and centrifuged within 30-45 min of collection, using a chemiluminescence technique (Immulite®2000TSH Third Generation).
Change from baseline in mean total HOMA-IR. | At baseline and week 12.
  The homeostasis model assessment (HOMA), an epidemiologic method for assessing insulin resistance [HOMA-IR=insulin (mU/ml) X glucose (mg/dl)/405] will be used as surrogate measure of insulin sensitivity
Change from baseline in mean total score of CES-D-R | At baseline and week 12.
  CESDR scale measure symptoms of depression in nine different groups as defined by the American Psychiatric Association Diagnostic and Statistical Manual, fifth edition. The Total CESD-R Score is calculated as a sum of responses to all 20 questions. The range of possible scores is between 0 (for those who say 'not at all or less than one day to all 20 questions' and 60 (for those who say '5-7 days' or 'nearly every day for 2 weeks' for all 20 questions). No clinical significance: a total CESD-R score less than 16 across all 20 questions.
Change from baseline in mean total score of Screen for Child Anxiety Related Emotional Disorders (SCARED). | At baseline and week 12.
  Appropriate screening tool to aid the diagnosis of anxiety disorders in adolescents attending an outpatient clinic.It consists of 41 items that are rated from 0 to 2, being 0 never, 1 sometimes and 2 always. The cut-off point is 25, that is, there is a probability of at least 70% that the child or adolescent has an anxiety disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Juárez de México, Mexico City, Mexico

REFERENCES:
- [Derived] Macias-Cortes E, Arellano-Alvarez S, Vega-Monroy S, Vera-Perez V, Llanes-Gonzalez L, Sanchez-Navarrete P, Enciso-Gonzalez D. Efficacy of Homeopathy in Addition to a Multidisciplinary Intervention for Overweight or Obesity in Mexican Adolescents: Study Protocol for a Randomized, Double-Blind, Placebo-Controlled Trial. Homeopathy. 2020 May;109(2):87-96. doi: 10.1055/s-0039-1697927. Epub 2020 Jan 20. PMID 31958867